CLINICAL TRIAL: NCT01502748
Title: Magnesium Therapy: a Novel Platform for Neuroprotectant Sampling in Acute Stroke
Brief Title: Endovascular Magnesium Sampling in Acute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: FAST-Mag study finished
Sponsor: University of Southern California (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, William Mack, Assistant Professor of Neurosurgery, University of Southern California
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS-11-00311; 12BGIA8700001 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2011-12-25; First posted 2012-01-02 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Acute Stroke
Keywords: stroke; Magnesium; Endovascular
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endovascular Sampling (Experimental): Paired sampling from the distal arterial(endovascular catheter) and peripheral venous (femoral sheath) locations in acute stroke patients undergoing endovascular recanalization who received intravenous Magnesium Sulfate as a part of the FAST-MAG study
  Interventions: Other: endovascular sampling

INTERVENTIONS:
Other: endovascular sampling — Paired sampling from the distal arterial(endovascular catheter) and peripheral venous (femoral sheath) locations: withdrawal of 3ml of blood from vasculature distal to the occlusive thrombus

SUMMARY:
This investigation will address the safety and feasibility of distal, intra-arterial sampling through endovascular access, in acute stroke patients. Levels of Magnesium will be measured in the region of infarct in patients who had been treated with intravenous Magnesium therapy following an acute stroke. This study attempts to address whether the traditional intravenous means of neuroprotectant administration achieves adequate concentration of the therapeutic agent in the area of diseased tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Patient with acute cerebral ischemia due to ICA or MCA occlusion,
2. Patient already enrolled in the NIH FAST-MAG clinical trial,
3. Patient's clinical attending physician plans mechanical embolectomy procedure as part of routine clinical care.
4. Age 40-95 inclusive (age criteria for FAST-MAG Trial).

Exclusion Criteria:

1. Technical inability to navigate microcatheter to target clot.
2. Patient or surrogate unavailable for consent

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Magnesium concentration | intra-procedure (at time of first pass of retrieval device)
  The primary endpoint is the relative concentration of Mg in the core cerebral ischemic zone, compared to systemic therapeutic Mg levels, as a measure of delivery efficacy of systemic administration.

SECONDARY OUTCOMES:
Sampling feasibility | intra-procedural (at time of first pass of retrieval device)
  sampling feasibility will be determined by the proportion of cases in which a cerebral circulation Mg level was successfully assayed
Safety | post-operative day 1
  safety will be assessed by intraoperative adverse events, postoperative neurologic examination including NIH stroke scale, and postoperative brain imaging.

CONTACTS AND LOCATIONS:
Overall Officials: William J Mack, MD, Principal Investigator — University of Southern California; Jeffrey Saver, MD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - University California Los Angeles: Ronald Reagan and Santa Monica Hospitals, Los Angeles, California
  - University of Southern California University and LA County Hospitals, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No